CLINICAL TRIAL: NCT02351869
Title: Nitrous Oxide as a Putative Novel Dual-Mechanism Treatment for Bipolar Disorder
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: This study was terminated due to COVID-19 pandemic-related halting of recruitment in the context of an upcoming replacement of the study MRI scanner.
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Principal Investigator, Dr. Benjamin Goldstein, Associate Professor, University of Toronto, Sunnybrook Health Sciences Centre
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 435-2013
Record Dates: First submitted 2014-12-02; First posted 2015-01-30 (Estimated); Last update posted 2023-04-06 (Actual); Status verified 2023-04

CONDITIONS: Bipolar Disorder
MeSH Terms: conditions — Bipolar Disorder | interventions — Nitrous Oxide; Midazolam

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Nitrous oxide (Active Comparator): N2O-condition participants will inhale an initial mixture of 10% N2O in oxygen (O2) for 5 minutes, followed by 25% N2O in O2 for 20 minutes. N2O-condition participants will also receive 5ml intravenous saline concomitantly with 10% N2O, and again with 25% N2O.
  Interventions: Drug: Nitrous Oxide
- Midazolam (Placebo Comparator): Inhaled room air plus intravenous midazolam bolus (total 2mg). Midazolam-condition participants will receive intravenous infusions of 0.5mg midazolam in 5ml saline (start of 1st inhalation epoch), followed by 1.5mg midazolam in 5ml saline (start of 2nd inhalation epoch).
  Interventions: Drug: Midazolam

INTERVENTIONS:
Drug: Nitrous Oxide
  Arms: Nitrous oxide
Drug: Midazolam
  Arms: Midazolam

SUMMARY:
This study is a 7-day randomized, double-blind proof-of-concept pilot study of nitrous oxide vs. midazolam in 40 adults (20-60 years) with bipolar disorder (BD) (type I or II). Ongoing pharmacological and psychosocial treatments may continue, provided that they have not been initiated or significantly modified in the preceding 2 weeks. Participants' current treatment as prescribed by clinical psychiatrists will not be modified or interfered in this study. The study involves 3 visits. During study visit 1, participants will complete screening to ensure study eligibility. This will be done using interview measures. During study visit 2, participants will complete anthropomorphic measurements, measurement of endothelial function, screening blood work, ECGs, and an anaesthesia screener. During study visit 3, participants will receive the treatment (nitrous oxide or midazolam), complete an MRI scan, and complete interview measures and self-reports. There will be anthropomorphic measurements taken as well. The participant will be required to complete phone interviews and self-reports over the subsequent 7 days. There are 4 main predictions: 1. Nitrous oxide will significantly reduce depression symptoms vs. midazolam. 2. Nitrous oxide will significantly increase frontal cortical perfusion vs. midazolam. 3. Lower perfusion in frontal cortical regions at baseline will be associated with greater improvement in depression symptoms following nitrous oxide treatment. 4. Poorer endothelial function will be associated with greater improvement in depression symptoms following nitrous oxide treatment.

ELIGIBILITY:
Inclusion Criteria:

English-speaking; age 20-60 years; BD-I or BD-II, current major depressive episode ≥4 weeks duration; MADRS≥22; taking ≥1 mood stabilizing medication/s (i.e. antimanic anticonvulsant, antipsychotic, and/or lithium).

Exclusion Criteria:

New medications or changes in dosing, or ECT or TMS, in the preceding 2 weeks; MADRS item 10, > 4; YMRS≥12; acute significant suicidality; psychosis; substance abuse (past 3 months); active major medical conditions (hepatic, renal, respiratory, or cardio/cerebrovascular disease; diabetes; esophageal reflux; sleep apnea); B12 deficiency/disorders; pregnant; MRI contraindications; history of adverse anaesthetic reactions; anaesthesia class >2; scuba diving in preceding week.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2015-08; Primary Completion 2020-02-01 (Actual); Study Completion 2020-06-07 (Actual)

PRIMARY OUTCOMES:
Change in Montgomery-Asberg Depression Scale (MADRS) score | Assessed at baseline, an average of 3 days later, again at up to 5 days after baseline on the day of drug administration, and participants will be followed for 7 days after the drug administration
  Measures mood symptom severity, used to select patients and assess treatment efficacy. Although other time-points will be examined, 24h was selected as the primary outcome to minimize the impact of acute sedation and psychoactive effects.

SECONDARY OUTCOMES:
Young Mania Rating Scale (YMRS) | Assessed at baseline, an average of 3 days later, again at up to 5 days after baseline on the day of drug administration, and participants will be followed for 7 days after the drug administration
  Measures symptom severity
Blood Pressure | Measured an average of 3 days post-baseline and again approximately every hour on the drug administration day
Weight | Assessed an average of 3 days after baseline
Beck Depression Inventory (BDI-II) | Assessed on the drug administration day and followed for 7 days post-drug administration
  Self-report measure of mood severity
Heart Rate | Measured an average of 3 days post-baseline and again approximately every hour on the drug administration day
Brief Psychiatric Rating Scale | Assessed on the drug administration day and followed for 7 days post-drug administration
The Clinician Administered Dissociative States Scale (CADSS) | Assessed on the drug administration day and followed for 7 days post-drug administration
General Information Sheet (Demographics) | Collected at baseline
  Demographics
Hamilton Anxiety Rating Scale (HAM-A) | Assessed on the drug administration day and followed for 7 days post-drug administration
  Interview measure used to assess anxiety severity
Hamilton Depression Rating Scale (HDRS) | Assessed on the drug administration day and followed for 7 days post-drug administration
  Interview measure used to assess mood severity
Patient Rated Inventory of Side Effects | Assessed on the drug administration day and followed for 7 days post-drug administration
  Self-report used to assess side effects
CANTAB Medication Listing | Assessed an average of 3 days after baseline
  Used to collect medications taken the day before and on the day of blood work
Structured Clinical Interview for DSM Disorders | Assessed at baseline
  Interview measure used to assess DSM disorders
Visual Analogue Scale | Assessed on the drug administration day and followed for 7 days post-drug administration
Height | Assessed an average of 3 days after baseline
Endothelial Function assessed via RH-PAT using the EndoPAT. | Assessed an average of 3 days after baseline and lasts approximately 30 minutes
  Will be assessed via RH-PAT using the EndoPAT.
Frontal Perfusion assessed using an MRI scan | Assessed approximately 5 days after baseline and post-drug administration
  Will be assessed using an MRI scan.
Biomarkers (B12 and nitric oxide (NO)) | Assessed an average of 3 days after baseline
  B12 and nitric oxide (NO) will be examined as predictors of response owing to known associations with the mechanism of action of N2O.

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin I Goldstein, MD, Principal Investigator — Sunnybrook Health Sciences Centre
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada

REFERENCES:
- [Result] Dimick MK, Omrin D, MacIntosh BJ, Mitchell RHB, Riegert D, Levitt A, Schaffer A, Belo S, Iazzetta J, Detzler G, Choi M, Choi S, Orser BA, Goldstein BI. Nitrous oxide as a putative novel dual-mechanism treatment for bipolar depression: Proof-of-concept study design and methodology. Contemp Clin Trials Commun. 2020 Jun 23;19:100600. doi: 10.1016/j.conctc.2020.100600. eCollection 2020 Sep. PMID 32637725
- [Result] Kim WSH, Dimick MK, Omrin D, Mitchell RHB, Riegert D, Levitt A, Schaffer A, Belo S, Iazzetta J, Detzler G, Choi M, Choi S, Herrmann N, McIntyre RS, MacIntosh BJ, Orser BA, Goldstein BI. Proof-of-concept randomized controlled trial of single-session nitrous oxide treatment for refractory bipolar depression: Focus on cerebrovascular target engagement. Bipolar Disord. 2023 May;25(3):221-232. doi: 10.1111/bdi.13288. Epub 2023 Jan 5. PMID 36579458